CLINICAL TRIAL: NCT04414839
Title: Comparison of Digital Intubation (Two-finger) and Video Laryngoscopy Methods During Nasogastric Tube Insertion in Intubated Patients
Brief Title: Comparison of Digital Intubation (Two-finger) and Video Laryngoscopy
Acronym: NGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Nasr Isfahani, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 397585
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Intubated Patients
Keywords: Digital Laryngoscopy; Endotracheal Tube; Nasogastric Tube (NGT); Video Laryngoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Intubation (Two-finger) (Active Comparator)
  Interventions: Device: Digital Intubation (Two-finger)
- Video Laryngoscopy (Active Comparator)
  Interventions: Device: Video Laryngoscopy

INTERVENTIONS:
Device: Digital Intubation (Two-finger) — In the NGT Digital Intubation group (group B), the second and third fingers were placed in the posterior pharynx and depressed the tongue downwards. The NGT was passed through the nose into the posterior pharynx with the fingers in the pharynx to reach the esophagus. The thumb was placed under the jaw and pushed it forward to pave the way for tube insertion.
  Arms: Digital Intubation (Two-finger)
Device: Video Laryngoscopy — In the NGT Video Laryngoscopy group (group A), first, the GlideScope blade was inserted under direct visualization via color monitor through the patient's mouth by employing jaw-thrust maneuver to preserve the cervical spine and by raising the tongue to obtain better visualization of the larynx space. Then, NGT was inserted through the selected nostril, advanced through the esophagus under direct vision to meet the measured length, and fixed after confirmation.
  Arms: Video Laryngoscopy

SUMMARY:
Abstract Background: A number of patients referring to the emergency departments (EDs) due to airway obstruction or decreased level of consciousness require the establishment of a definite airway using intubation. On the other hand, performing Nasogastric tube (NGT) insertion is very challenging in anesthetized and intubated patients. And, a conclusive method has not yet been presented in this regard. Hence, the current study aimed at comparing Digital Intubation (two-finger) and Video Laryngoscopy methods during NGT insertion.

Materials and Methods: The present clinical trial was performed on 76 intubated patients that were randomly divided into two groups. Groups A and B underwent Video Laryngoscopy and Digital Intubation (two-finger) methods, respectively. Then, the success rate, the number of attempts to insert NGT, duration of insertion, hemodynamic parameters, and patients' satisfaction level were recorded and examined in this study.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year old patients that underwent rapid sequence intubation (RSI) and required NGT insertion

Exclusion Criteria:

* having skull base fracture symptoms
* coagulopathy and hemorrhagic disorders
* maxillofacial traumas leading to the deformity and disturbance in NGT insertion
* diseases and anomalies of the upper respiratory tract
* deviated nasal septum
* nostril stenosis
* esophageal disorders (esophageal stricture, esophageal varices)
* a history of head and neck radiotherapy, and
* patients intubated in and transferred from other centers
* patients with more than two unsuccessful attempts at NGT insertion were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Success rate | Procedure (The start time was when NGT entered the selected nostril, and the end time was when the measured NGT length was fully entered the stomach.)
  being successfully inserted into the stomach

SECONDARY OUTCOMES:
Insertion duration | Procedure (The start time was when NGT entered the selected nostril, and the end time was when the measured NGT length was fully entered the stomach.)
  Measuring how long will it last to insert successfully an NG tube into the stomach

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahra University Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided
if requested, it will be shared formally by email to the journal office.